CLINICAL TRIAL: NCT04781218
Title: ABC Science Collaborative Registry Study
Status: Withdrawn | Type: Observational
Why Stopped: Study did not start
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00107036
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-03

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants enrolled in the registry: Participants enrolled in the registry will include school community members including students, parents, staff, etc.

SUMMARY:
The ABC Registry is associated with Pro00107943 and provides a resource for collecting information on members of school communities both regionally in North and South Carolina, as well as nationally in the United States (U.S.) through the National Program, including children, parents, teachers, superintendents, and other staff; and children identified through clinical practice. The overall goals of the Registry are to collect data relevant to public health during the coronavirus 2019 (COVID-19) pandemic and to establish and engage school communities that may be eligible for participation in future research studies, including observational studies, as well as prospective COVID-19 trials.

ELIGIBILITY:
Inclusion Criteria:

* Participant currently attends, is the parent of a student, works in, or works with a school that is participating in the ABC Science Collaborative, or participant is an adult or child who learned of the registry through clinical practice and is interested in participating in COVID-19 related research,
* Participant or their parent/guardian has provided informed consent or assent, as applicable
* Participant or their parent/guardian has downloaded the "ABC Science" App from the App store as a part of the ABC Science Collaborative and has agreed to the App's Terms of Use
* Participant or their parent/guardian is able to speak and read English or Spanish

Exclusion Criteria:

* There are no specific exclusion criteria for this registry. Participants must meet inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: School community members, including students, parents, staff, etc.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Participants who enroll in the ABC Registry | Up to 5 years
  Number of participants who enroll in the ABC Registry (e.g. are interested in participating in upcoming research studies, including those related to COVID-19).

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://abcsciencecollaborative.org/